CLINICAL TRIAL: NCT01084590
Title: Healthy Homes/Healthy Kids: Pediatric Primary Care-based Obesity Prevention
Brief Title: Healthy Homes/Healthy Kids_5-9
Acronym: HHHK_5-9
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Washington (Other); University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A08-132; 1R01DK084475 (NIH)
Record Dates: First submitted 2010-03-09; First posted 2010-03-10 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Obesity; Injury
Keywords: Prevention; Obesity; Safety; Unhealthy weight gain; Injury prevention
MeSH Terms: conditions — Obesity; Wounds and Injuries | interventions — Diet, Healthy; Exercise; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy Eating/Physical Activity (Experimental): This intervention arm will include brief pediatrician counseling regarding the child's current BMI percentile status, recommendations for home environmental changes to achieve a healthy weight gain trajectory, and home safety and injury risk reduction environmental recommendations paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the obesity prevention home environmental strategies.
  Interventions: Behavioral: Healthy Eating/Physical Activity
- Safety/Injury Prevention (Active Comparator): This intervention arm will include the same brief counseling from the pediatrician paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the safety and injury prevention home environmental strategies.
  Interventions: Behavioral: Safety/Injury Prevention

INTERVENTIONS:
Behavioral: Healthy Eating/Physical Activity — This intervention arm will include brief pediatrician counseling regarding the child's current BMI percentile status, recommendations for home environmental changes to achieve a healthy weight gain trajectory, and home safety and injury risk reduction environmental recommendations paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the obesity prevention home environmental strategies.
  Arms: Healthy Eating/Physical Activity
Behavioral: Safety/Injury Prevention — This intervention arm will include the same brief counseling from the pediatrician paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the safety and injury prevention home environmental strategies.
  Arms: Safety/Injury Prevention

SUMMARY:
The pediatric primary care setting is a relatively untapped resource for addressing obesity prevention. The main goal of this study is to evaluate the efficacy of a relatively low cost pediatric primary-care based obesity prevention intervention. The intervention will consist of brief pediatrician counseling as well as phone coaching for parents with overweight children who are between the ages of five and nine. We propose to enroll and randomize 425 parent-child dyads with children who have a measured body mass index (BMI) the 75th and 95th percentile. They will be randomized one of into two groups, the (a) Healthy Eating/Physical Activity Intervention, or the (b) General Healthy/Safety/Injury Prevention Contact Control Intervention. Both groups will receive brief pediatrician counseling regarding their child's current BMI percentile status and recommendations for home environmental changes to achieve a healthy weight gain trajectory and to improve home safety and reduce injury risk. This will be paired with a 12 month home-based program delivered via phone by health behavior specialists to help parents make environmental changes specific to their group assignment.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the efficacy of a relatively low cost pediatric primary-care based intervention that integrates brief pediatric counseling and a home-based phone program to prevent unhealthy weight gain in overweight children ages five-nine. Parent-child dyads will be recruited for the Healthy Homes/Healthy Kids Study via a multi-step process including use of electronic medical record data to identify children, pediatrician approval, and outreach via letters and phone calls. Four hundred and twenty five parent-child dyads from pediatric primary care will be recruited to participate and be randomized to one of two interventions:

Healthy Eating/Physical Activity Home-based Intervention: This intervention arm will include brief pediatrician counseling regarding the child's current BMI percentile status, recommendations for home environmental changes to achieve a healthy weight gain trajectory, and home safety and injury risk reduction environmental recommendations paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the obesity prevention home environmental strategies.

Safety/Injury Prevention Home-based Contact Control Intervention: This intervention arm will include the same brief counseling from the pediatrician paired with a 12 month home-based program delivered via phone by a masters-level health behavior specialist to promote implementation of the safety and injury prevention home environmental strategies.

ELIGIBILITY:
Inclusion Criteria:

* BMI%ile between the 75th and 95th%ile
* Receives care at a HealthPartners Clinic in the Twin Cities Metropolitan Area

Exclusion Criteria:

* Children with the following chronic conditions: kidney disease, Type 1 diabetes, lupus, a thyroid condition, cancer, or chromosomal abnormality such as Down's syndrome or Turner's syndrome
* Children who within the last six months or those who are currently taking the following medications and took them or will be taking them for more than a month: Prednisone, Prednisilone, and Decadron.
* Families who have limited English skills.
* Families who plan to move out of the metropolitan area within the next two years.

Ages: 5 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 421 (Actual)
Dates: Start 2010-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
BMI percentile change | 24 months
  Children at risk for obesity (defined as having a BMI%ile between the 75th and 85th%ile) whose parent participates in the Healthy Eating/Physical Activity Intervention will have a significantly lower BMI percentile at 12 and 24 month-follow up when compared to children whose parents participated in the Safety/Injury Prevention Intervention.

SECONDARY OUTCOMES:
Dietary intake and activity patterns | 24 months
  Children whose parents are in the Healthy Eating/Physical Activity Home-based Intervention participants will exhibit more favorable dietary intake and activity patterns relative to children whose parents are in the Safety/Injury Prevention group
Parenting behaviors | 24 months
  Parents who exhibit more parenting behaviors related to obesity prevention and higher overall adherence to pediatric primary care provider recommendations will be more successful in helping their child achieve a healthy weight gain trajectory.
BMI percentile and psychosocial adjustment | 24 months
  A lower increase in BMI percentile will be associated with more favorable psychosocial adjustment and that there will be no increase in disordered eating in children with parents in the Healthy Eating/Physical Activity group relative to children with parents in in the Safety/Injury Prevention group
Parent BMI | 24 months
  Parent attention to child weight and instruction to model healthy eating and physical activity behavior will impact parent weight, with the Healthy Eating/Physical Activity group parents having lower BMI relative to the Safety/Injury Prevention group parents.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy E Sherwood, PhD, Principal Investigator — HealthPartners Institute; Rona L Levy, PhD, Principal Investigator — University of Washington School of Social Work
Locations (2):
- United States (2):
  - HealthPartners Research Foundation, Bloomington, Minnesota
  - University of Washington School of Social Work, Seattle, Washington

REFERENCES:
- [Derived] JaKa MM, French SA, Wolfson J, Jeffery RW, Lorencatto F, Michie S, Levy RL, Langer SL, Sherwood NE. Understanding Outcomes in Behavior Change Interventions to Prevent Pediatric Obesity: The Role of Dose and Behavior Change Techniques. Health Educ Behav. 2019 Apr;46(2):312-321. doi: 10.1177/1090198118798679. Epub 2018 Sep 14. PMID 30215279
- [Derived] Kunin-Batson AS, Seburg EM, Crain AL, Jaka MM, Langer SL, Levy RL, Sherwood NE. Household factors, family behavior patterns, and adherence to dietary and physical activity guidelines among children at risk for obesity. J Nutr Educ Behav. 2015 May-Jun;47(3):206-15. doi: 10.1016/j.jneb.2015.01.002. Epub 2015 Mar 4. PMID 25748634
- [Derived] Sherwood NE, Levy RL, Langer SL, Senso MM, Crain AL, Hayes MG, Anderson JD, Seburg EM, Jeffery RW. Healthy Homes/Healthy Kids: a randomized trial of a pediatric primary care-based obesity prevention intervention for at-risk 5-10 year olds. Contemp Clin Trials. 2013 Sep;36(1):228-43. doi: 10.1016/j.cct.2013.06.017. Epub 2013 Jun 28. PMID 23816490